CLINICAL TRIAL: NCT02906917
Title: This Trial is Conducted Globally. The Aim of This Trial is to Compare the Effect and Safety of Insulin Degludec/Insulin Aspart vs. Insulin Glargine Plus Insulin Aspart in Subjects With Type 2 Diabetes Treated With Basal Insulin With or Without Oral Antidiabetic Treatment in Need of Treatment Intensification.
Brief Title: A 38 Week Trial Comparing Effect and Safety of Insulin Degludec/Insulin Aspart vs. Insulin Glargine Plus Insulin Aspart in Subjects With Type 2 Diabetes Treated With Basal Insulin With or Without Oral Antidiabetic Treatment in Need of Treatment Intensification
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-4266; 2015-004768-12 (EudraCT Number); U1111-1175-7895 (Other: WHO)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDegAsp (Experimental)
  Interventions: Drug: Insulin degludec/insulin aspart
- IGlar + IAsp (Active Comparator)
  Interventions: Drug: Insulin glargine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin degludec/insulin aspart — Administered subcutaneously (s.c. under the skin) once daily.
  Arms: IDegAsp
Drug: Insulin glargine — Administered subcutaneously (s.c. under the skin) once daily.
  Arms: IGlar + IAsp
Drug: Insulin aspart — Administered subcutaneously (s.c. under the skin) once daily.
  Arms: IGlar + IAsp

SUMMARY:
Trial comparing effect and safety of insulin degludec/insulin aspart vs. insulin glargine plus insulin aspart in subjects with type 2 diabetes treated with basal insulin with or without oral antidiabetic treatment in need of treatment intensification.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age at least 18 years at the time of signing informed consent Algeria: Male or female, age at least 19 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus
* Treated with any basal insulin for at least 90 days prior to the day of screening
* Subject not on any OAD(s) prior to trial participation OR subjects on stable daily dose(s) of OAD(s) for at least 90 days prior to screening visit (V1). The OAD(s) include any of the following anti-diabetic drug s)/regimen: a. Biguanides (metformin at least 1500 mg or maximum tolerated dose documented in the subject medical record) b. Other OADs (at least half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record): i. Insulin secretagogues (SU and glinides) ii. Di-peptidyl-peptidase IV (DPP-4) inhibitors iii. α-glucosidase inhibitors iv. Sodium/glucose co-transporter 2 (SGLT-2) inhibitors v. Oral combination products (of the allowed individual OADs above)
* HbA1c 7.0-10.0% (53-86 mmol/mol) (both inclusive) by central laboratory analysis
* Body mass index (BMI) equal to or below 45.0 kg/m^2

Exclusion Criteria:

* Participation in any clinical trial of an approved or non-approved investigational medicinal product within four weeks prior to the day of screening (V1)
* Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent severe metabolic dysregulation (e.g. diabetes ketoacidosis) equal or below 90 days prior to the day of the screening and between screening and randomisation
* Any of the following: myocardial infarction, stroke or hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and between screening and randomisation
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of below 60 ml/min/1.73 m^2 as defined by KDIGO 2012 classification using isotope dilution mass spectrometry (IDMS) for serum creatinine measured at screening
* Impaired liver function, defined as alanine aminotransferase (ALT) equal to or above 2.5 times upper normal limit (UNL) at screening.
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (58):
- United States (29):
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Danbury, Connecticut
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Westfield, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Bartlett, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
- Algeria (3):
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sidi Bel Abbes
- Czechia (4):
  - Novo Nordisk Investigational Site, Broumov
  - Novo Nordisk Investigational Site, Náchod
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Trutnov
- India (9):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Surat, Gujarat
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Aurangabad, Maharashtra
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Russia (7):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Cheboksary
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Syktyvkar
  - Novo Nordisk Investigational Site, Tyumen
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir

REFERENCES:
- [Result] Philis-Tsimikas A, Astamirova K, Gupta Y, Haggag A, Roula D, Bak BA, Fita EG, Nielsen AM, Demir T. Similar glycaemic control with less nocturnal hypoglycaemia in a 38-week trial comparing the IDegAsp co-formulation with insulin glargine U100 and insulin aspart in basal insulin-treated subjects with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2019 Jan;147:157-165. doi: 10.1016/j.diabres.2018.10.024. Epub 2018 Nov 16. PMID 30448451
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 71 sites in 7 countries, as follows: Algeria (4), Czech Republic (6), India (10), Russian Federation (11), Serbia (5), Turkey (7), and United States (28). Additionally, 1 site in the United States screened, but didn't randomise any subject.
Groups:
- Insulin Degludec/Insulin Aspart: Subjects received treatment for 38 weeks as per the following sequence: 1) Initiation period (period-1, week 0-26): Insulin degludec/insulin aspart (IDegAsp) once daily (OD) administered at the largest meal each day with or without oral antidiabetic drug(s) (OAD(s)). Subjects switching from pre-trial basal insulin OD or more to IDegAsp OD at trial entry were to transfer unit-to-unit. 2) Intensification period (period-2, week 26-38): IDegAsp OD/twice a day (BID) administered at the largest meal(s) each day (in the case of BID dosing, one meal being dinner) based on individual needs with or without OAD(s).
- Insulin Glargine + Insulin Aspart: Subjects received treatment for 38 weeks as per the following sequence: 1) Initiation period (period-1, week 0-26): Insulin glargine (IGlar) OD administered in accordance with local labelling and insulin aspart (IAsp) OD administered at the largest meal with or without OAD(s). Subjects switching from pre-trial basal insulin OD to IGlar OD were also to transfer unit-to-unit to IGlar, while subjects switching from basal insulin more than OD to IGlar OD were to reduce the initial total daily dose by 20% or according to local labelling. IAsp was to be initiated at 4 units with the largest meal. 2) Intensification period (period-2, week 26-38): IGlar OD administered in accordance with local labelling and IAsp 1-3 times daily administered at main meals based on individual needs with or without OAD(s).
Period: Initiation Period (Week 0-26)
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Started | 267 | 265
Exposed | 265 | 263
Completed | 261 | 254
Not Completed | 6 | 11
Not completed — Unclassified | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 3 | 4
Period: Intensification Period (Week 26-38)
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Started | 261 | 254
Completed | 252 | 247
Not Completed | 9 | 7
Not completed — Unclassified | 3 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), which included all randomised subjects.
Groups:
- Insulin Degludec/Insulin Aspart: Subjects received treatment for 38 weeks as per the following sequence: 1) Initiation period (period-1, week 0-26): IDegAsp OD administered at the largest meal each day with or without OAD(s). Subjects switching from pre-trial basal insulin OD or more to IDegAsp OD at trial entry were to transfer unit-to-unit. 2) Intensification period (period-2, week 26-38): IDegAsp OD/BID administered at the largest meal(s) each day (in the case of BID dosing, one meal being dinner) based on individual needs with or without OAD(s).
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart | Total
Number analyzed (Participants) | 267 | 265 | 532
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (8.9) | 59.2 (9.1) | 58.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 128 | 270
  Male | 125 | 137 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 41
  Not Hispanic or Latino | 246 | 245 | 491
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 29 | 32 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 221 | 220 | 441
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (%) - Week 26
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated 26 weeks after randomisation.
Time Frame: Week 0, week 26
Population: FAS, which included all randomised subjects. Number of subjects analyzed = number of subjects contributed to the analysis at specified time point.
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
% of HbA1c
  Baseline (week 0): number analyzed (Participants) | 261 | 264
  Baseline (week 0) | 8.2 (0.8) | 8.1 (0.7)
  Change from baseline (week 26): number analyzed (Participants) | 251 | 248
  Change from baseline (week 26) | -1.1 (0.9) | -1.1 (0.8)
Statistical Analysis 1: Comparison: Insulin Degludec/Insulin Aspart vs Insulin Glargine + Insulin Aspart; The response and change from baseline in response are analysed on 1000 complete, imputed data sets after multiple imputation for each treatment arm separately. A penalty of 0.4% is added to the week 26 values for all premature treatment discontinued subjects, and subject with missing HbA1c values at week 26 in the IDegAsp arm. Each of the imputed data sets are analysed through an analysis of covariance (ANCOVA); Test type: Non-Inferiority — Non-inferiority of IDegAsp OD versus IGlar OD + IAsp OD was considered confirmed if the 95% confidence interval for the mean treatment difference was entirely below 0.40%; p < 0.0001, ANCOVA — One-sided p-value for test of non-inferiority; Treatment, region, sex, previous insulin treatment and previous OAD treatment as categorical fixed effects and baseline response and age as covariate; Treatment contrast = 0.07, 95% CI 2-sided [-0.06 to 0.21]

2. Secondary Outcome: Change in HbA1c (%) - Week 38
Description: Change from baseline (week 0) in HbA1c was evaluated 38 weeks after randomisation.
Time Frame: Week 0, week 38
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
% of HbA1c
  Baseline (week 0): number analyzed (Participants) | 261 | 264
  Baseline (week 0) | 8.2 (0.8) | 8.1 (0.7)
  Change from baseline (week 38): number analyzed (Participants) | 247 | 242
  Change from baseline (week 38) | -1.2 (0.9) | -1.2 (0.9)

3. Secondary Outcome: Responder (Yes/No) for HbA1c < 7%
Description: Participants achieving (yes/no) HbA1c <7% was evaluated 26 and 38 weeks after randomisation, respectively.
Time Frame: Week 26 and week 38
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
Number of participants
  Week 26: Yes: number analyzed (Participants) | 241 | 242
  Week 26: Yes | 120 | 120
  Week 26: No: number analyzed (Participants) | 241 | 242
  Week 26: No | 121 | 122
  Week 38: Yes: number analyzed (Participants) | 234 | 233
  Week 38: Yes | 139 | 140
  Week 38: No: number analyzed (Participants) | 234 | 233
  Week 38: No | 95 | 93

4. Secondary Outcome: Responder (Yes/No) for HbA1c <7% Without Severe or BG Confirmed Symptomatic Hypoglycaemia
Description: Participants achieving (yes/no) HbA1c <7% without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia, was evaluated 26 and 38 weeks after randomisation, respectively. Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Severe hypoglycaemia as per ADA classification: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: Week 26 and week 38
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
Number of participants
  Week 26: Yes: number analyzed (Participants) | 241 | 242
  Week 26: Yes | 73 | 61
  Week 26: No: number analyzed (Participants) | 241 | 242
  Week 26: No | 168 | 181
  Week 38: Yes: number analyzed (Participants) | 234 | 233
  Week 38: Yes | 60 | 56
  Week 38: No: number analyzed (Participants) | 234 | 233
  Week 38: No | 174 | 177

5. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated 26 and 38 weeks after randomisation, respectively.
Time Frame: Week 0, week 26, week 38
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
mg/dL
  Baseline: Week 0: number analyzed (Participants) | 257 | 261
  Baseline: Week 0 | 162.4 (47.8) | 157.8 (47.8)
  Change from baseline: Week 26: number analyzed (Participants) | 231 | 231
  Change from baseline: Week 26 | -42.1 (52.1) | -40.6 (59.2)
  Change from baseline: Week 38: number analyzed (Participants) | 225 | 230
  Change from baseline: Week 38 | -48.6 (54.2) | -41.5 (55.3)

6. Secondary Outcome: Change in Pre-breakfast SMPG (Used for Titration)
Description: Reported results are observed pre-breakfast self-measured plasma glucose (SMPG; used for titration) values at week 1 (baseline) and 26 and 38 weeks after randomisation.
Time Frame: Week 1, week 26, week 38
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
mg/dL
  Week 1 (Baseline): number analyzed (Participants) | 264 | 259
  Week 1 (Baseline) | 158.3 (45.7) | 149.4 (43.8)
  Week 26: number analyzed (Participants) | 242 | 243
  Week 26 | 107.5 (24.8) | 103.4 (20.7)
  Week 38: number analyzed (Participants) | 235 | 234
  Week 38 | 102.9 (20.0) | 103.8 (22.5)

7. Secondary Outcome: Change in Postprandial SMPG Increment (From 9-point Profile)
Description: Change from baseline (week 0) in postprandial SMPG increment (from 9-point profile) was evaluated 26 and 38 weeks after randomisation, respectively. 9-point SMPG profiles were measured starting in the morning 2 days prior to the scheduled visit at the time points described below: 1) Before breakfast (2 days prior to visit) 2) 90 minutes after start of the breakfast 3) Before lunch 4) 90 minutes after start of the lunch 5) Before dinner/main evening meal 6) 90 minutes after start of the dinner/main evening meal 7) At bedtime (2 days or 1 day prior to visit depending on actual clock time) 8) At 4 a.m. (1 day prior to visit) 9) Before breakfast at the following day (1 day prior to the visit).
Time Frame: Week 0, week 26, week 38
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 267 | 265
mg/dL
  Baseline: Week 0: number analyzed (Participants) | 264 | 261
  Baseline: Week 0 | 54.5 (37.7) | 48.4 (38.0)
  Change from baseline: Week 26: number analyzed (Participants) | 234 | 240
  Change from baseline: Week 26 | -10.8 (46.3) | -8.7 (40.6)
  Change from baseline: Week 38: number analyzed (Participants) | 224 | 221
  Change from baseline: Week 38 | -17.7 (40.0) | -19.7 (45.0)

8. Secondary Outcome: Number of Nocturnal, Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of nocturnal, treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were analysed during the following periods: weeks 0-26, weeks 16-26 and weeks 0-38. Nocturnal hypoglycaemic episodes: episodes occurring between 00:01 and 05:59 both inclusive. Treatment emergent: hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product.
Time Frame: Weeks 0-26, weeks 16-26, weeks 0-38
Population: Safety analysis set, which included all subjects receiving at least one dose of the investigational product (IDegAsp) or comparator (IGlar). Number of subjects analyzed = number of subjects contributed to the analysis at specified time point.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 265 | 263
Episodes
  Weeks 0-26 | 61 | 118
  Weeks 16-26: number analyzed (Participants) | 251 | 250
  Weeks 16-26 | 24 | 58
  Weeks 0-38 | 113 | 189

9. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were analysed during the following periods: weeks 0-26, weeks 16-26 and weeks 0-38. Treatment emergent: hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product.
Time Frame: Weeks 0-26, weeks 16-26, weeks 0-38
Population: Safety analysis set, which included all subjects receiving at least one dose of the investigational product or comparator. Number of subjects analyzed = number of subjects contributed to the analysis at specified time point.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 265 | 263
Episodes
  Weeks 0-26 | 329 | 376
  Weeks 16-26: number analyzed (Participants) | 251 | 250
  Weeks 16-26 | 154 | 194
  Weeks 0-38 | 537 | 640

10. Secondary Outcome: Total Insulin Dose
Description: Total insulin dose was evaluated 26 and 38 weeks after randomisation, respectively.
Time Frame: Week 26 and week 38
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 265 | 263
Units
  Week 26: number analyzed (Participants) | 242 | 243
  Week 26 | 70.9 (41.5) | 79.4 (37.7)
  Week 38: number analyzed (Participants) | 235 | 234
  Week 38 | 83.4 (51.3) | 89.3 (43.1)

11. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated 26 and 38 weeks after randomisation, respectively.
Time Frame: Week 0, week 26, week 38
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 265 | 263
Kg
  Baseline: Week 0 | 88.5 (18.6) | 88.4 (17.5)
  Change from basline: Week 26: number analyzed (Participants) | 242 | 242
  Change from basline: Week 26 | 1.7 (3.2) | 1.4 (3.2)
  Change from basline: Week 38: number analyzed (Participants) | 235 | 235
  Change from basline: Week 38 | 2.5 (3.8) | 2.4 (3.2)

12. Secondary Outcome: Incidence of TEAEs
Description: Number of treatment emergent adverse events (TEAEs) were analysed during the following periods: weeks 0-26, weeks 26-38 and weeks 0-38. Treatment emergent: An adverse event that had an onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. If an event had an onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period, or if it had an onset date within 7 days after the last drug date, then this event was also to be considered as a TEAE.
Time Frame: Weeks 0-26, weeks 26-38, weeks 0-38
Population: as for outcome 8
Measure: Number; unit: Events
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
Number analyzed (Participants) | 265 | 263
Events
  Weeks 0-26 | 441 | 408
  Weeks 26-38: number analyzed (Participants) | 245 | 243
  Weeks 26-38 | 173 | 117
  Weeks 0-38 | 614 | 525

ADVERSE EVENTS:
Time Frame: Week 0 to week 38 (treatment period) + 7 days (follow-up period).
Description: All presented adverse events are treatment emergent (i.e., TEAEs). Results are based on the safety analysis set, which included all subjects receiving at least one dose of the investigational product.
Arm/Group | Insulin Degludec/Insulin Aspart | Insulin Glargine + Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 0/265 | 2/263
Serious Adverse Events (participants affected / at risk) | 18/265 | 20/263
Other Adverse Events (participants affected / at risk) | 74/265 | 57/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Insulin Aspart (N=265) | Insulin Glargine + Insulin Aspart (N=263)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Insulin Aspart (N=265) | Insulin Glargine + Insulin Aspart (N=263)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 9 (9)
Headache (Nervous system disorders) | 27 (52) | 16 (23)
Nasopharyngitis (Infections and infestations) | 36 (49) | 22 (27)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02906917/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02906917/SAP_001.pdf